CLINICAL TRIAL: NCT02306031
Title: The Effect of Topical Sodium Diclofenac on Macular Thickness in Diabetic Eyes After Phacoemulsification: A Randomized Controlled Trial
Brief Title: Topical Diclofenac on Macular Thickness After Phacoemulsification
Acronym: diclofenac
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88108
Record Dates: First submitted 2014-11-15; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Diabetic Oculopathy
Keywords: diclofenac; macular thickness; phacoemulsification; OCT(Optical coherence tomography ); diabetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (ARTIFICIAL TEAR) (Placebo Comparator): control group received artificial tear (Sina Darou Laboratories Company, Tehran, Iran) as a placebo every 6 hours. Theses drops continued up to 6 weeks with the same dose after operations.
  Interventions: Drug: Prescribe ARTIFICIAL TEAR
- diclofenac sodium drop (Active Comparator): case group received diclofenac sodium drop 0.1% (Sina Darou Laboratories Company, Tehran, Iran) every 6 hours.. Theses drops continued up to 6 weeks with the same dose after operations.
  Interventions: Drug: Prescribe diclofenac sodium drop 0.1%

INTERVENTIONS:
Drug: Prescribe ARTIFICIAL TEAR — From one week before surgery, and control group received artificial tear (Sina Darou Laboratories Company, Tehran, Iran) as a placebo every 6 hours. Theses drops continued up to 6 weeks with the same dose after operations
  Arms: placebo (ARTIFICIAL TEAR)
Drug: Prescribe diclofenac sodium drop 0.1% — From one week before surgery, case group received diclofenac sodium drop 0.1% (Sina Darou Laboratories Company, Tehran, Iran) every 6 hours.Theses drops continued up to 6 weeks with the same dose after operations
  Arms: diclofenac sodium drop

SUMMARY:
Eyes of 108 diabetic patients have underwent phacoemulsification and intraocular lens implantation surgery have enrolled. Fifty four eyes have received the conventional postoperative care with steroid drop, whereas the other group (54 eyes) have given a preoperative diclofenac drop four times daily in addition to steroid drop and continued six weeks after surgery. All patients have evaluated by Optical coherence tomography (OCT) preoperatively and days 1, 30, and 90.The outcome measures including best corrected visual acuity (BCVA) and OCT findings were compared in and between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with non-proliferative diabetic retinopathy that were candidate for phacoemulsification and intraocular lens implantation

Exclusion Criteria:

* Eyes with clinically significant macular edema based on the ETDRS(Early Treatment Diabetic Retinopathy Study) study and/or central macular thickness >260µ were not included. Neither did we include the eyes with other accompanying diseases affecting the macula or eyes with history of previous retinal laser photocoagulation or intraocular surgery.
* Eyes with severe cataract that preclude performing an acceptable quality optical coherence tomography (OCT) were not enrolled either.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
macular thickness changes | preoperatively until 90 days
  Optical coherence tomography (OCT)

SECONDARY OUTCOMES:
best corrected visual acuity (BCVA) changes | preoperatively until 90 days
  LogMAR (Logarithm of the Minimum Angle of Resolution)charts

CONTACTS AND LOCATIONS:
Locations (1):
- Labbafinejad medical center, Tehran, Iran